CLINICAL TRIAL: NCT00788970
Title: Shiatsu Adjuvant Therapy And Placebo For Schizophrenia:a Double Blind Study
Brief Title: Shiatsu Adjuvant Therapy And Placebo For Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Herzog Hospital (Other)
Responsible Party: Dr. Pesach Lichtenberg, Herzog Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: lichtenberg3
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia
Keywords: Acupressure; Shiatsu; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupressure (Experimental): Acupressure adjuvant therapy
  Interventions: Behavioral: Acupressure adjuvant therapy
- Placebo acupressure (Placebo Comparator): Sham acupressure adjuvant therapy
  Interventions: Behavioral: Acupressure adjuvant therapy
- No treatment (No Intervention): Wait list group (no treatment)

INTERVENTIONS:
Behavioral: Acupressure adjuvant therapy — Acupressure provided in 40-minute sessions, twice a week for 4 weeks. For placebo acupressure, different meridian points will be used.
  Other Names: Shiatsu
  Arms: Acupressure; Placebo acupressure

SUMMARY:
In the current study we will study the effect of adding acupressure (shiatsu) to conventional therapy in treating individuals with schizophrenia.

DETAILED DESCRIPTION:
Acupressure, also known as shiatsu, is a holistic form of medicine originating in Japan but now widely practiced throughout the world. The theory is based on Traditional Chinese Medicine (TCM), which sees meridians of life force (chi) running through the body, and aims to optimize health through manipulating the body into maximal alignment.

We are proposing a randomized double-blind placebo-controlled trial to examine the efficacy of acupressure as adjuvant therapy added to antipsychotics in the treatment of patients with schizophrenia.

The goals of this study are twofold:

1. To assess through the highest standards of empirical research whether acupressure can benefit patients with schizophrenia.
2. To furnish data relevant to the possible physiological mechanisms by which acupressure may produce a therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV diagnosis of schizophrenia or schizoaffective disorder
2. Ages 18 and over
3. Clinical status stable, as reflected by changes in Brief Psychiatric Rating Scale (BPRS) (Overall & Gorham, 1961) of less than 20% during a one month period prior to randomization, and at least one month of drug treatment without change of anti-psychotic drug or dosage.
4. Ability to cooperate with 40-minute sessions

Exclusion Criteria:

1. Unstable general medical conditions
2. Active bone fracture or other orthopedic problem
3. Skin condition that renders treatment unsafe or painful
4. Active infection in skin or soft tissues, such as cellulitis
5. Solid tissue malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Lichtenberg, M.D., Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Department of Psychiatry, Jerusalem, Israel